CLINICAL TRIAL: NCT06164808
Title: Cardiac Arrhythmia Telemetry; Conventional vs HeartWatch
Acronym: CATCH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HelpWear Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CATCH V1.0
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Cardiac Arrhythmia; Diagnostic/Monitoring Devices Related to Adverse Incidents
MeSH Terms: conditions — Arrhythmias, Cardiac; Disease

STUDY DESIGN:
Intervention Model Description: All subjects will wear the Holter monitor and the HeartWatch.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active device engagement (Other): All subjects will wear either the Holter monitor and the HeartWatch.
  Interventions: Device: HeartWatch

INTERVENTIONS:
Device: HeartWatch — The HeartWatch is indicated for the extended diagnostic evaluation of patients with symptomatic and transient symptoms such as light-headedness, syncope, and palpitations, as well as patients at risk for arrhythmias, but without significant symptoms. It is an armband consisting of the main body of the device with an additional sensor located on the band. It is worn around the upper left arm to obtain heart electrical signals. The device is paired with the HelpWear application on a smartphone where the signals are stored and then will be uploaded to a secure network for analysis.

SUMMARY:
Heart rhythm disorders are common and significantly impact the lives of those affected and their families. The main problems can be categorized as: a) atrial fibrillation or AF and atrial flutter, b) supra-ventricular tachycardia or SVT, c) excessively slow heart beats (i.e., bradycardia or pauses) and d) ventricular arrhythmias. These problems can be difficult to detect with currently available monitoring options as they are all worn for shorter terms or are an invasive implantable option. The HeartWatch is a longer term monitoring system that is worn on the upper arm, allows users to create a tag and pairs with an app on a smartphone allowing for correlation of symptoms.

DETAILED DESCRIPTION:
Patients who are being referred to wear a holter monitor will be approached to wear a HeartWatch simultaneously. This will allow collection of signals on both devices and to compare the accuracy of signals between the Heartwatch vs Holter monitor. It will also examine the reliability of autodetect algorythms between the devices. We will also collect information to compare the amount of adverse events between the various systems and the patient preference of those systems.

ELIGIBILITY:
Inclusion Criteria:

* At least 22 years of age at time of consent
* Clinically indicated for a Holter monitor test
* Able to wear the HeartWatch on the left bicep for the study duration
* Able to follow the protocol
* No functional implantable pacemaker or defibrillator
* Left bicep circumference >/= 22 cm and </= 45 cm
* Provision of written-informed consent

Exclusion Criteria:

* Known allergy to any component of the Holter monitor
* Known allergy to any component of the HeartWatch
* Inability to wear the HeartWatch on the left arm for the study period due to pre-existing medical condition (3.g., functional AV fistula in left arm, prior carcinoma with lymph node dissection or lymphedema, known blood clot of recurrent blood clots in the left arm, chronic neuropathic pain in left arm, ...)
* Dextrocardia
* Implanted functional Pacemaker or Defibrillator
* Left bicep circumference < 22 cm
* Left bicep circumference < 45 cm

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
QRS signal detection | For the duration of time that the patient wears the Holter monitor and the HeartWatch, 24-48 hours
  Compare QRS detection accuracy with HeartWatch data vs. the Holter monitor lead I signal

SECONDARY OUTCOMES:
ECG strip evaluation | For the duration of time that the subject wears the holter vs the HeartWatch (24-48 hours).
  Compare the overall agreement of the HeartWatch vs. Holter data in providing interpretable ECG strips data for all symptomatic (patient tagged) events and all cardiologist-verified non-normal rhythms identified by cardiology technologists (Holter).
ECG PR interval assessment | For the duration of time that the subject wears the holter vs the HeartWatch (24-48 hours).
  Assess the comparability of paired, 10-minute averaged PR intervals measured from the HeartWatch vs. the Holter lead I reference signal.
ECG QRS interval assessment | For the duration of time that the subject wears the holter vs the HeartWatch (24-48 hours).
  Assess the comparability of paired, 10-minute averaged QRS intervals measured from the HeartWatch vs. the Holter lead I reference signal.
ECG interval assessment | For the duration of time that the subject wears the holter vs the HeartWatch (24-48 hours).
  Assess the comparability of paired, 10-minute averaged heart rate corrected QT (QTc) intervals measured from the HeartWatch vs. the Holter lead I reference signal.

OTHER OUTCOMES:
Adverse events | For the duration of time that the subject wears the holter vs the HeartWatch (24-48 hours).
  Evaluate and describe adverse events related to the use of the HeartWatch and Holter devices.
User preference | For the duration of time that the subject wears the holter vs the HeartWatch (24-48 hours).
  Compare user preferences for the HeartWatch and Holter devices
ECG strip categorization | For the duration of time that the patient wears the Holter monitor and the HeartWatch, 24-48 hours.
  Compare ECG strip categorizations of the HeartWatch vs. the Holter.
Future software validation | Data obtained during the recordings will be used for future software validation for 5 years.
  To use the ECG data signals collected to validate future software

CONTACTS AND LOCATIONS:
Overall Officials: Russell Quinn, MD, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No